CLINICAL TRIAL: NCT03680599
Title: Connection to Health for Smokers -- A Comprehensive Program to Reduce Tobacco-Related Health Disparities in CHCs
Brief Title: Connection to Health for Smokers
Acronym: CTHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27IP-0024
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connection to Health for Smokers (Experimental): Participants in this arm will participate in the Connection to Health for Smokers Arm of the study, wherein an electronic survey will be administered and participants will be guided through an evidence-based action planning sequence, taking into account each patient's unique social environment, health related behaviors, and behavioral health status, with multimodal follow up.
  Interventions: Behavioral: Connection to Health for Smokers
- Enhanced Standard of Care (Active Comparator): Participants in this arm will participate in Enhanced Standard Care, wherein participants will receive a brief electronic survey and receive standard smoking cessation program that does not include formal action planning and multimodal follow up.
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Connection to Health for Smokers — Connection to Health for Smokers includes 5 core components supported by online tools: (1) comprehensive electronic patient survey, (2) automated summary report to flag areas of difficulty (3) interactive priority setting, (4) interactive action planning, and (5) electronic text reminders and followup.
  Arms: Connection to Health for Smokers
Behavioral: Enhanced Standard of Care — Participants will complete a survey and receive standard one-on-one smoking cessation according to a usual care protocol delivered by health educators
  Arms: Enhanced Standard of Care

SUMMARY:
The goal of the study is to develop and test Connection to Health for Smokers (CTHS), a comprehensive program to support smokers to quit and improve smokers' general health. The program will be designed for implementation by health educators in community health centers.

DETAILED DESCRIPTION:
The investigators will use a participatory approach to develop and test the feasibility and acceptability of CTHS in community health center sites in Contra Costa County. Development of the program will be informed by active engagement with a patient advisory group composed of current smokers and clinical team members who serve current smokers in community health centers. Feasibility and acceptability will be assessed by implementing the CTHS program for patients in 3 clinical sites, using the RE-AIM evaluation framework. Primary outcomes will include the number and proportion of enrolled smokers who create at least one health-related action plan with a health educator, and stated intention of clinical teams to continue using CTHS after the research. The investigators will enroll 90 smokers in CTHS and 90 additional smokers in Enhanced Standard of Care (ESC) which will be the active comparison group. Participants will be randomly assigned. Smoking status will be reassessed after 3 months. Primary outcomes will include number of 24-hour quit attempts, and 7-day smoking abstinence, as well as changes in self-efficacy and readiness to quit smoking among participants who do not quit. Results of this pilot program will inform further development of the CTHS program for testing in larger scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

- Must have smoked cigarettes in the last 7 days

Exclusion Criteria:

- Speaking languages other than English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Program Reach, Effectiveness, Adoption, Implementation, and Maintenance | 3 months
  The RE-AIM Framework will be used to assess program feasibility

SECONDARY OUTCOMES:
7-day smoking abstinence | 3 months
  Not smoking cigarettes (not even a puff) in the last 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Potter, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No